CLINICAL TRIAL: NCT03302923
Title: Effects of Brisk Walking on Autonomic Nervous System Reactivation in Nursing Home Residents.
Brief Title: Brisk Walking Study in Nursing Home Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Mutualiste Chirurgicale de la Loire (Other)
Collaborators: University Hospital of Saint-Etienne (Other); University of Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08; 2016-A00068-43 (Registry Identifier: ANSM)
Record Dates: First submitted 2017-09-28; First posted 2017-10-05 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Physical Activity; Autonomic Nervous System Imbalance
Keywords: Nursing home residents; Brisk walking
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brisk walking 1 (Experimental): 1 time a week of 9 months brisk walking
  Interventions: Behavioral: Brisk walking
- Brisk walking 3 (Experimental): 3 times a week of 9 months brisk walking
  Interventions: Behavioral: Brisk walking
- Control group (No Intervention): No brisk walking session

INTERVENTIONS:
Behavioral: Brisk walking — Prospective randomized clinical trial with 2 intervention groups and 1 control group.
  Arms: Brisk walking 1; Brisk walking 3

SUMMARY:
It is well established that physical activity reduces the physiological effects of ageing. Among them, the decrease of the autonomic nervous system activity (ANS) is associated with the increase of cardiovascular events and sleep disorders occurence. It has been shown that high intensity cycle training can enhance the ANS activity by 30% in people aged of 70 years old. However, such trainings were done by old athletes used to train at intensities that could not be handled by nursing home elderly. Thus, an adapted activity such as brisk walking shall be defined to make it practicable for the many in convalescent homes. The investigators hypothesize that long term brisk walking training could lead to reactivate ANS in people living in convalescent homes.

DETAILED DESCRIPTION:
The investigators aim to compare the effects of a 9 month brisk walking training (1 time a week or 3 times a week) on the ANS of nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* Being over 60 years old
* Living in a nursing home of Mutualité Française de la Loire, France
* Being able to walk without human aid
* Being able to speak and write French
* Being inactive (less than 1 hours of physical activity per week)
* Having a normal sinus rhythm
* Being affiliated to the social welfare system
* Signing the informed consent form

Exclusion Criteria:

* Having serious balance disorders
* Suffering from cardiac or respiratory pathologies that contraindicate physical activity
* Serious comorbidities contraindicating physical activity
* Diagnosed cardiac pathologies that prevent heart rate variability analysis: congestive heart failure, cardiac pacemaker, implantable cardioverter defibrillator, serious ventricular rhythm troubles, atrial fibrillation, atrial flutter.
* Persons under legal protection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
SDNN value | 9 months
  Standard deviation of all normal nocturnal RR intervals

SECONDARY OUTCOMES:
Heart rate variability parameters | 9 months
  Autonomic nervous system balance (RMSSD)
Heart rate variability parameters | 9 months
  Autonomic nervous system balance (LF/HF)
Heart rate variability parameters | 9 months
  Autonomic nervous system balance (Ptot)
Baroreflex sensitivity (BRS) | 9 months
  BRS slope variation measured at rest
Maximum oxygen uptake (VO2max) | 9 months
  Cardiopulmonary exercise testing
Daily physical activity | 9 months
  Actimetry (Actigraph-GT3X)
Daily physical activity | 9 months
  Adult physical activity questionnaire (APAQ)
Sedentary periods | 9 months
  Actimetry (Actigraph GT3X)
Sedentary periods | 9 months
  Adult physical activity questionnaire (APAQ)
Muscular force | 9 months
  Lower limbs maximum voluntary force test measured on force chair
Muscular endurance | 9 months
  Lower limbs endurance test measured on force chair
Muscular volume gains | 9 months
  Lower limbs muscular magnetic resonance imaging (MRI)
Plasmatic dosages of inflammatory molecules | 9 months
  CRP
Plasmatic dosages of inflammatory molecules | 9 months
  TNF alpha
Plasmatic dosages of inflammatory molecules | 9 months
  IL 17
Cognitive improvements | 9 months
  Neuropsychological evaluation with a neuropsychologist.
Quality of life | 9 months
  SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, PhD, Principal Investigator — University Hospital of Saint-Etienne
Locations (1):
- French Loire Mutuality, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No